CLINICAL TRIAL: NCT05709977
Title: Acupuncture for Nasal Congestion in Allergic Rhinitis: An Open-Label, Randomized, Monocenter Trial (ANCAR Trial)
Brief Title: Acupuncture for Nasal Congestion in Allergic Rhinitis
Acronym: ANCAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johanna Maria Vermeulen (Other)
Collaborators: Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Mermaid Medicine® (Other)
Responsible Party: Sponsor-Investigator, Johanna Maria Vermeulen, Principal Investigator, Mermaid Medicine®
Organization: Mermaid Medicine® (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANCAR Trial
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Allergic Rhinitis
Keywords: Acupuncture; Nasal Congestion; Allergic Rhinitis; Randomized
MeSH Terms: conditions — Rhinitis, Allergic; Nasal Obstruction | interventions — Acupuncture Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized, Controlled, Interventional, Monocenter Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture arm (Experimental): Fixed set of acupuncture points
  Interventions: Other: Acupuncture
- Control (Carelastin®) arm (Active Comparator): Carelastin® (1 mg/ml) azelastine nasal spray, 1 spray puff (0.14 ml) per nostril twice daily (totally 0.56 ml per day)
  Interventions: Drug: Antihistamine nasal spray

INTERVENTIONS:
Other: Acupuncture — Fixed set of acupuncture points
  Arms: Acupuncture arm
Drug: Antihistamine nasal spray — Carelastin® (1 mg/ml) azelastine nasal spray
  Other Names: Intranasal antihistamine (INAH) therapy
  Arms: Control (Carelastin®) arm

SUMMARY:
Allergic rhinitis (AR) is a disorder that affects more than 500 million people worldwide. Nasal congestion is one of the most general and bothersome symptoms in rhinitis, which affects the quality of life (QOL). Current medications are undesirable due to their side-effects. Acupuncture for AR in general can be considered as safe and can be seen as a potential therapeutic intervention for nasal congestion. Evidence supported that acupuncture is clinically used for signs and symptoms of nose disorders, such as nasal congestion, with effectiveness, but whether acupuncture has immediate, post-treatment and long-term effects on nasal congestion in AR is not verified by strictly designed clinical study. The ANCAR trial uses a standard treatment protocol with a fixed set of acupuncture points - to be as scientific as possible from Western medical viewpoint - to open the nose and affect underlying energetic imbalance and immunity at the same time, to maintain its nose opening effect. This novel acupuncture treatment protocol can be seen as a solid and profound approach from which every AR patient may benefit.

DETAILED DESCRIPTION:
Worldwide more than approximately 500 million people suffer from AR (30% of the Dutch population) and its prevalence is expanding. Nasal congestion (i.e. reversible mucosal congestion/nasal mucosal obstruction) is one of the most general and bothersome symptoms in rhinitis and is associated with other medical conditions such as rhinosinusitis and otitis media. This study is relevant as in addition to the high global occurrence of AR, this disorder has substantial effects on the quality of life (QOL) (e.g. during sleep and work). AR is related to high direct medical costs (mainly prescription of medications and outpatient visits) and indirect economic costs (including productivity decrease). Current medications are undesirable due to their side-effects (such as sedation in the case of intranasal antihistamines (INAH)).

Acupuncture for AR in general can be considered as safe and can be seen as a potential therapeutic intervention for nasal congestion. Evidence supported that acupuncture is clinically used for signs and symptoms of nose disorders, such as nasal congestion, with effectiveness, but whether acupuncture has immediate, post-treatment and long-term effects on specifically nasal congestion in AR is not verified by strictly designed clinical study. The ANCAR trial aims to evaluate the effects of an acupuncture treatment protocol for nasal congestion in AR compare to azelastine nasal spray (Carelastin®). A standard treatment protocol with a fixed set of acupuncture points has been established - to be as scientific as possible from Western medical viewpoint - and this selection of acupuncture points can be seen as a solid and profound approach from which every AR patient may benefit. This standard set opens the nose and affects the underlying energetic imbalance and immunity at the same time to maintain its nose opening effect (i.e. to prevent recurrence of the complaint). The acupuncture protocol concerns 8 treatments during 6 weeks (i.e. 2 treatments per week during the first 2 weeks and 1 treatment per week in the consecutive 4 weeks).

The positive effects of this treatment protocol (such as improvement QOL) may result in more confidence in the direct, post-treatment and long-term effects of acupuncture and lead to more acceptance of acupuncture as a solid treatment option for nasal congestion in AR instead of using an INAH spray.

Hypothesis: Acupuncture will improve nasal congestion in AR compare to azelastine nasal spray (Carelastin®).

Objective: To evaluate the effects of an acupuncture treatment protocol for nasal congestion in AR.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed AR by a physician
* Have one of the AR types: seasonal (SAR) or perennial (PAR) or mixed (MAR) allergic rhinitis
* VAS nasal congestion: 3-10
* Age: from 18 years
* Signed Informed Consent

Exclusion Criteria:

* COVID-19
* Acute common cold
* Influenza
* Fever (38°C or higher)
* Acute nasal trauma (such as a fracture and epistaxis)
* Irreversible nasal blockages (such as septum deviation, concha bullosa, polyps and cysts)
* Nasal and sinus cancer
* Pregnancy or planning for pregnancy
* Consumed decongestions, antihistamines, antibiotics or corticosteroids within 2 weeks before the RCT
* Received acupuncture, Chinese herbal medicine or another complementary treatment within 2 weeks before the RCT
* Received immunotherapy within 2 weeks before the RCT
* Participants refusing or unable to sign Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | After 6 weeks (visit 8).
  To compare the effects of acupuncture and azelastine nasal spray (Carelastin®) on nasal congestion in AR after 6 weeks of treatments based on VAS score. VAS, 0 = no nasal congestion, and 10 = most severe nasal congestion.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | At 1st day (visit 1), During 6 weeks of treatments (visit 2-7: Only acupuncture arm), 2 weeks after treatment protocol (visit 9), and 2 months after treatment protocol (visit 10).
  To compare the effects of acupuncture and azelastine nasal spray (Carelastin®) on nasal congestion in AR after different visits of treatments based on VAS score. VAS, 0 = no nasal congestion, and 10 = most severe nasal congestion.
Peak Nasal Inspiratory Flow (PNIF) | At 1st day (visit 1), After 6 weeks (visit 8), 2 weeks after treatment protocol (visit 9), and 2 months after treatment protocol (visit 10).
  To compare the effects of acupuncture and azelastine nasal spray (Carelastin®) on nasal congestion in AR after different visits of treatments based on PNIF score (score ranges between 30-370 L/min).
Adapted Nasal Obstruction Symptom Evaluation (NOSE) | After 6 weeks (visit 8), and 2 months after treatment protocol (visit 10).
  To compare the effects of acupuncture and azelastine nasal spray (Carelastin®) on nasal congestion in AR after different visits of treatments based on Adapted NOSE score. NOSE, 0 = no problem, and 4 = severe problem.
Visual Analog Scale (VAS) | At 1st day (visit 1), During 6 weeks of treatments (visit 2-7: Only acupuncture arm), After 6 weeks (visit 8), 2 weeks after treatment protocol (visit 9), and 2 months after treatment protocol (visit 10).
  To assess the effects of acupuncture on other nasal and ocular signs and symptoms in AR based on VAS score. VAS, 0 = no symptom, and 10 = most severe symptom.
Adapted Nasal Obstruction Symptom Evaluation (NOSE) | After 6 weeks (visit 8), and 2 months after treatment protocol (visit 10).
  To assess the effects of acupuncture on general health, concentration and energy level in AR after different visits of treatments based on Adapted NOSE score. NOSE, 0 = excellent, and 4 = poor.
Adapted Nasal Obstruction Symptom Evaluation (NOSE) | After 6 weeks (visit 8), and 2 months after treatment protocol (visit 10).
  To assess the effects of acupuncture on equalization of middle ear pressure in AR in the case patients fly and/or dive after different visits of treatments based on adapted NOSE score. NOSE, 0 = no problem, 4 = severe problem, and 99 = not applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna M. Vermeulen, BSc., L.Ac., Principal Investigator — Mermaid Medicine®
Locations (1):
- Mermaid Medicine®, The Hague, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlies the results reported in this article after deidentification (text, tables, figures and appendixes) for qualified researchers. Approval of the request is a prerequisite to the sharing of data.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 months following publication, ending 3 years following article publication.
Access Criteria: Access to trial IPD can be requested by a qualified researcher engaging in independent scientific research.
URL: https://www.mermaidmedicine.com

REFERENCES:
- [Background] Bousquet J, Khaltaev N, Cruz AA, Denburg J, Fokkens WJ, Togias A, Zuberbier T, Baena-Cagnani CE, Canonica GW, van Weel C, Agache I, Ait-Khaled N, Bachert C, Blaiss MS, Bonini S, Boulet LP, Bousquet PJ, Camargos P, Carlsen KH, Chen Y, Custovic A, Dahl R, Demoly P, Douagui H, Durham SR, van Wijk RG, Kalayci O, Kaliner MA, Kim YY, Kowalski ML, Kuna P, Le LT, Lemiere C, Li J, Lockey RF, Mavale-Manuel S, Meltzer EO, Mohammad Y, Mullol J, Naclerio R, O'Hehir RE, Ohta K, Ouedraogo S, Palkonen S, Papadopoulos N, Passalacqua G, Pawankar R, Popov TA, Rabe KF, Rosado-Pinto J, Scadding GK, Simons FE, Toskala E, Valovirta E, van Cauwenberge P, Wang DY, Wickman M, Yawn BP, Yorgancioglu A, Yusuf OM, Zar H, Annesi-Maesano I, Bateman ED, Ben Kheder A, Boakye DA, Bouchard J, Burney P, Busse WW, Chan-Yeung M, Chavannes NH, Chuchalin A, Dolen WK, Emuzyte R, Grouse L, Humbert M, Jackson C, Johnston SL, Keith PK, Kemp JP, Klossek JM, Larenas-Linnemann D, Lipworth B, Malo JL, Marshall GD, Naspitz C, Nekam K, Niggemann B, Nizankowska-Mogilnicka E, Okamoto Y, Orru MP, Potter P, Price D, Stoloff SW, Vandenplas O, Viegi G, Williams D; World Health Organization; GA(2)LEN; AllerGen. Allergic Rhinitis and its Impact on Asthma (ARIA) 2008 update (in collaboration with the World Health Organization, GA(2)LEN and AllerGen). Allergy. 2008 Apr;63 Suppl 86:8-160. doi: 10.1111/j.1398-9995.2007.01620.x. No abstract available. PMID 18331513
- [Background] Kjaergaard T, Cvancarova M, Steinsvag SK. Nasal congestion index: A measure for nasal obstruction. Laryngoscope. 2009 Aug;119(8):1628-32. doi: 10.1002/lary.20505. PMID 19507219
- [Background] Ichimura K. Mechanism of nasal obstruction in patients with allergic rhinitis. Clin Exp Allergy. 2010;10(1):20-27. https://doi.org/10.1111/j.1472-9733.2010.01151.x.
- [Background] Lieberman P, Kaliner MA, Wheeler WJ. Open-label evaluation of azelastine nasal spray in patients with seasonal allergic rhinitis and nonallergic vasomotor rhinitis. Curr Med Res Opin. 2005 Apr;21(4):611-8. doi: 10.1185/030079905X41408. PMID 15899111
- [Background] Craig TJ, Sherkat A, Safaee S. Congestion and sleep impairment in allergic rhinitis. Curr Allergy Asthma Rep. 2010 Mar;10(2):113-21. doi: 10.1007/s11882-010-0091-5. PMID 20425503
- [Background] Skoner DP. Complications of allergic rhinitis. J Allergy Clin Immunol. 2000 Jun;105(6 Pt 2):S605-9. doi: 10.1067/mai.2000.106150. PMID 10856165
- [Background] Bousquet PJ, Demoly P, Devillier P, Mesbah K, Bousquet J. Impact of allergic rhinitis symptoms on quality of life in primary care. Int Arch Allergy Immunol. 2013;160(4):393-400. doi: 10.1159/000342991. Epub 2012 Nov 23. PMID 23183377
- [Background] Law AW, Reed SD, Sundy JS, Schulman KA. Direct costs of allergic rhinitis in the United States: estimates from the 1996 Medical Expenditure Panel Survey. J Allergy Clin Immunol. 2003 Feb;111(2):296-300. doi: 10.1067/mai.2003.68. PMID 12589348
- [Background] Wallace DV, Dykewicz MS, Bernstein DI, Blessing-Moore J, Cox L, Khan DA, Lang DM, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CC, Schuller D, Spector SL, Tilles SA; Joint Task Force on Practice; American Academy of Allergy; Asthma & Immunology; American College of Allergy; Asthma and Immunology; Joint Council of Allergy, Asthma and Immunology. The diagnosis and management of rhinitis: an updated practice parameter. J Allergy Clin Immunol. 2008 Aug;122(2 Suppl):S1-84. doi: 10.1016/j.jaci.2008.06.003. No abstract available. PMID 18662584
- [Background] Sertel S, Bergmann Z, Ratzlaff K, Baumann I, Greten HJ, Plinkert PK. Acupuncture for nasal congestion: a prospective, randomized, double-blind, placebo-controlled clinical pilot study. Am J Rhinol Allergy. 2009 Nov-Dec;23(6):e23-8. doi: 10.2500/ajra.2009.23.3380. Epub 2009 Sep 18. PMID 19769799
- See also: Mylan website. Allergische rhinitis. Updated November 13, 2018. Accessed December 3, 2021. Website inactive on March 13, 2024. — https://www.mylan.nl/nl-nl/therapeutische-gebieden/allergische-rhinitis